CLINICAL TRIAL: NCT00741442
Title: Randomized, Double-Blind, Multicenter,Placebo-Controlled, Dose Ranging, Efficacy and Safety Study of RDEA806 in Hyperuricemic Subjects With Symptomatic Gout
Brief Title: A Study of RDEA806 in Hyperuricemic Subjects With Symptomatic Gout
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RDEA806-501
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-01

CONDITIONS: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): RDEA806 400 mg qd
  Interventions: Drug: RDEA806
- 3 (Experimental): RDEA806 400 mg bid
  Interventions: Drug: RDEA806
- 2 (Placebo Comparator): Placebo QD
  Interventions: Drug: Placebo
- 4 (Placebo Comparator): Placebo BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RDEA806 — Uricosuric agent for the treatment of gout
  Arms: 1; 3
Drug: Placebo — Matching Placebo.
  Arms: 2; 4

SUMMARY:
The purpose of this study is to determine whether RDEA806 is effective in the treatment of hyperuricemia in gout patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient is hyperuricemic: screening serum uric acid ≥8 mg/dL.
* Patient meets one or more of the 1977 ARA criteria for the diagnosis of gout.
* Patient is willing and able to give informed consent and adhere to visit/protocol schedules
* All female subjects of child-bearing potential must agree to use a barrier method of birth control (e.g. condom, diaphragm or cap).

Exclusion Criteria:

* Consumes more than 14 drinks of alcohol per week.
* History or suspicion of drug abuse.
* History of kidney stones, rheumatoid arthritis or other autoimmune disease, significant cardiac dysfunction.
* Diabetes Mellitus requiring treatment
* Confirmed or suspected HIV-1 infection.
* Malignancy, except treated non-melanomatous skin cancer and cervical dysplasia.
* Uncontrolled hypertension.
* Inadequate renal function.
* Hemoglobin < 8 g/dL (males) or < 7 g/dL (females).
* ALT, AST , or GGT 2 x ULN
* Active peptic ulcer disease.
* Requires long-term use of salicylates; thiazide diuretics; losartan; azathioprine; mercaptopurine; theophylline; IV colchicine; cyclosporine; cyclophosphamide; pyrazinamide; sulfamethoxazole; trimethoprim.
* Pregnant or breast feeding.
* Use of an investigational drug within 4 weeks prior to study drug administration.
* Known hypersensitivity or allergy to RDEA806 or colchicine or any components in their formulations.
* Any other medical or psychological condition which, in the opinion of the investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements, or to complete the study.
* History of cardiac abnormalities including abnormal and clinically relevant ECG changes.
* Conditions predisposing to QT prolongation.
* Any use of concomitant medications that prolong the QT/QTc interval within 14 days prior to Day 1.
* Subjects with a QTcF interval >450 milliseconds at screening or on Day -1 or at pre-dose (Hour 0) on Day 1.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-07; Primary Completion 2009-04 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To compare the proportion of subjects whose serum uric acid (sUA) level is <6.0 mg/dL following 4 weeks of continuous treatment with RDEA806. | 4 weeks

SECONDARY OUTCOMES:
To evaluate the proportion of subjects whose sUA levels are <6.0 mg/dL, <5.0 mg/dL and <4.0 mg/dL, at each visit. | 4 weeks
To evaluate the absolute and percent reduction from baseline in sUA levels | 4 weeks
To evaluate percent change in 24-hour urine uric acid level | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Hingorani, MD, PhD, MBA, Study Director — Ardea Biosciences, Inc.
Locations (1):
- Toronto, Ontario, Canada